CLINICAL TRIAL: NCT04016129
Title: CART Immunotherapy Targeting CD19 Negative Acute Lymphoblastic Leukemia
Brief Title: CAR-T Immunotherapy Targeting CD19- ALL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-19003
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: B-cell Leukemia
Keywords: CD19- B-ALL; CART; CD22, CD123, CD38, CD10, CD20, TSLPR
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR-CD22/CD123/CD38/CD10/CD20/TSLPR (Experimental): Patients who have relapsed after CD19 CART immunotherapy or have CD19 negative B cell malignancies
  Interventions: Biological: 4SCAR-CD22/CD123/CD38/CD10/CD20/TSLPR

INTERVENTIONS:
Biological: 4SCAR-CD22/CD123/CD38/CD10/CD20/TSLPR — 4SCAR-CD22/CD123/CD38/CD10/CD20/TSLPR Patients who have relapsed after CD19 CART immunotherapy or have CD19 negative B cell malignancies

SUMMARY:
This study will evaluate safety and efficacy of a combination of 4th generation chimeric antigen receptor gene-modified T cells targeting CD19 negative ALL that express CD22, CD123, CD38, CD10, CD20 and TSLPR, as many patients developed CD19-negative disease after CD19 CART immunotherapy. Clinical response and development of a standardized lentiviral vector and cell production protocol will be investigated. This is a phase I/II trial enrolling patients from multiple clinical centers.

DETAILED DESCRIPTION:
Anti-CD19 chimeric antigen receptor T cell therapy has demonstrated unprecedented treatment responses in relapsing/refractory B-cell acute lymphoblastic leukemia (r/r B-ALL). However, many studies have reported that a subset of patients still relapse and about 30-50% of those relapses are characterized by the loss of CD19 surface antigen. Patients with CD19-negative relapse after CD19 CAR-T-cell therapy usually have a poor prognosis. The mechanisms underlying CD19-negative relapses are not fully understood and it is important to develop solutions to supplement post-CD19 immunotherapies.

Potential markers for recurrent leukemic blasts in an emerging CD19-negative blast population include many known B-cell lineage antigens. To prevent further target escape and improve the therapeutic effects, CAR gene-modified T cells targeting CD22, CD123, CD38, CD10, CD20 or TSLPR have been considered in post CD19 CAR-T immunotherapy. This study aims to evaluate safety and efficacy of administrating one or multiple non-CD19 targeting CAR-T cells to patients with CD19-negative B cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Native CD19 negative B cell malignancies or relapse after CD19-CAR-T immunotherapy.
3. Malignant B cells expressing one or more of the following surface molecules: CD22/CD123/CD38/CD10/CD20/TSLPR.
4. The KPS score over 80 points, and survival time is more than 1 month.
5. Greater than Hgb 80 g/L.
6. No contraindications to blood cell collection.

Exclusion Criteria:

1. Complications with other active diseases, and difficult to assess patient response.
2. Bacteria, fungus, or virus infection, and unable to control.
3. Living with HIV.
4. Active HBV and HCV infection.
5. Pregnant and nursing mothers.
6. Under systemic steroid use within a week of the treatment.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion | 24 weeks
  Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Anti-tumor activity of CART | 1 year
  Scale of CAR copies are detected by qPCR and leukemic cell burden are assessed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (3):
- China (3):
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Zhongxi Children Hospital, Shijiazhuang, Hebei